CLINICAL TRIAL: NCT00136344
Title: Antibiotic Prophylaxis for Cataract Surgery Version 7e January 22 2003
Brief Title: Study of Antibiotic Prophylaxis for Endophthalmitis Following Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: The European Society of Cataract and Refractive Surgeons(ESCRS) (Unknown); Santen Gmbh (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: MREC Ref. no. 02/5/46
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2007-06

CONDITIONS: Endophthalmitis
Keywords: cataract surgery; phacoemulsification; post-operative endophthalmitis
MeSH Terms: conditions — Endophthalmitis | interventions — Cefuroxime; Levofloxacin

INTERVENTIONS:
Drug: Cefuroxime
Drug: Levofloxacin

SUMMARY:
Cataract is the most important cause of visual impairment and decreased mobility in the elderly. While surgery is usually successful, it is also responsible for permanent loss of vision in up to 0.1% of patients due to severe post-operative infection (endophthalmitis). Because of this risk, surgery is typically performed on one eye at a time leaving the patient with a monocular cataract causing considerable visual impairment with reduction in mobility and quality of life. A second operation is required which often takes place up to one year later.

It is not known at present whether the post-operative complication of endophthalmitis can be prevented by perioperative use of antibiotics. This randomised study (masked and placebo-controlled for topical levofloxacin and unmasked for intracameral injection of cefuroxime) sets out to test in 4 groups, each of 8,750 cataract surgery patients, if either topical antibiotic (levofloxacin) perioperatively or an intraocular (intracameral) injection of antibiotic (cefuroxime) at the end of phacoemulsification cataract surgery or the combination provides effective prophylaxis of post-operative infection (endophthalmitis) compared to controls in whom perioperative antibiotics are not used. The result will provide a scientific basis for prophylaxis of infection (endophthalmitis) following cataract surgery in Europe as well as an accurate figure for the incidence of endophthalmitis following phacoemulsification cataract surgery in Europe for the first time.

DETAILED DESCRIPTION:
Cataract extraction with intra-ocular lens implantation is the most commonly performed surgical procedure in the elderly population in Europe. The frequency varies in different European Union (EU) countries involving 2 to 7 per 1000 population per annum. A population with an ever-increasing proportion of the elderly is advancing this figure with numbers requiring surgery expected to increase by 70% by 2006. While technical advances (phacoemulsification) have enhanced the efficacy of the procedure, the possibility of serious post-operative infection with loss of vision remains the most important unsolved problem.

In the absence of scientific evidence, the European Society of Cataract and Refractive Surgeons (ESCRS) wishes to determine whether one currently developed method of delivering antibiotics intraocularly in Sweden is of benefit compared to surgery without the use of perioperative antibiotics, as currently practised in many European centres, or to the use of frequent application of topical antibiotic drops perioperatively. The ESCRS also wishes to assess possible risk factors for later endophthalmitis.

This study requires four groups of 8,750 patients - 35,000 in all - to demonstrate reductions of currently reported rates of endophthalmitis (approximately 0.3%) in patients where no intraocular antibiotics are used, or where they are used by the subconjunctival route. Other studies using intraocular vancomycin have reported results as low as 0.05%, but these studies were not standardised or controlled and the results were anecdotal. In addition, vancomycin should not be used for routine prophylaxis and should only be used as the antibiotic of 'last resort'.

This multi-centre randomised study involves 24 operating units in 8 EU countries (Austria, Belgium, England, Germany, Italy, Poland, Portugal and Spain) and Turkey. Results in 8,750 patients receiving an intracameral injection of antibiotic (cefuroxime) at the end of surgery will be compared to 8,750 patients receiving topical antibiotic (levofloxacin) prophylaxis before and at the end of surgery, 8,750 patients receiving the combination and 8,750 patients receiving neither regime; in addition, all patients will receive povidone iodine antiseptic prophylaxis prior to surgery and post-operative levofloxacin from days 1 to 6 to prevent wound infection.

This group size will be sufficiently large to ensure at least 80% statistical power to detect a reduction of incidence from 0.25% to 0.08% using 5% significance level tests.

Surgical data from all patients will be collected directly into computers based within each operating theatre and transmitted to a central server in Glasgow (University of Strathclyde). Follow-up data for the presence or absence of endophthalmitis will be collected from all patients at post-operative visits and similarly recorded on computers for transmission to the central server. Sophisticated techniques will be used to check all data as it is uploaded.

ELIGIBILITY:
Inclusion Criteria:

* All patients, including diabetics, undergoing routine cataract surgery in each unit taking part in the study

Exclusion Criteria:

* Patients who do not wish to take part in the trial
* Patients allergic to penicillins and cephalosporins.
* Long-term nursing home patients
* Patients with only one eye
* Pregnancy.
* Children less than 18 years old.
* All severely 'at-risk' groups for infection including:

  * Severe atopic keratoconjunctivitis;
  * Severe active blepharitis;
  * Ocular cicatricial pemphigoid.
* Patients with complicated cataracts such as traumatic or subluxated
* Patients having combined operations with cataract surgery such as trabeculectomy or a corneal graft.
* Patients known to be allergic to povidone iodine (very rare) or any other known hypersensitivity to any components of the study medications.
* Patients who are incapacitated mentally and incapable of giving consent.
* Patients with severe thyroid disease
* Open infection anywhere, infection of lacrimal drainage channels or infection around the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35000
Dates: Start 2003-09; Study Completion 2006-05

PRIMARY OUTCOMES:
Prevention of post-operative endophthalmitis following phacoemulsification cataract surgery in Europe due to use of perioperative antibiotics
Incidence of endophthalmitis in Europe following phacoemulsification cataract surgery

SECONDARY OUTCOMES:
Effect of risk factors on the presentation of endophthalmitis in Europe following phacoemulsification cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter Barry, FRCS, Study Chair — ESCRS (European Society of Cataract and Refractive Surgeons); Mary D'Ardis, Principal Investigator — ESCRS
Locations (24):
- University Eye Clinic, Paracelsus Private Medical University, Salzburg, Austria
- Belgium (5):
  - University Hospital Antwerp, UZA Ophthalmology, Antwerp
  - University of Gent, Universitaire Zeikenhuis, Ghent
  - Jan Yperman Ziekenhuis, Ieper
  - Centre Hospitalier Universitaire, Liège
  - Oogheelkunde, Melveren
- Augenklinik Ahaus, Ahaus, Germany
- Italy (2):
  - Azienda Ospedaliera di Desenzano del Garda, Desenzano
  - Ospedale Borgo Trento, Verona
- Kierownik Katedry i Kliniki, Warsaw, Poland
- University Hospital, Coimbra, Portugal
- Spain (4):
  - Instituto Oftalmologico VISSUM, Alicante
  - La Candelaria University Hospital, La Candelaria, Tenerife
  - Hospital Universitario de Canarias, La Laguna, Tenerife
  - Hospital Oftalmologico Internacional, Madrid
- Dokuz Eylul University, Izmir, Turkey (Türkiye)
- United Kingdom (8):
  - Axminster Hospital, Axminster
  - West of England Eye Unit, Royal Devon & Exeter Hospital (Wonford), Exeter
  - Ipswich Hospital, Ipswich
  - Moorfields Eye Outreach Unit, Northwick Park Hospital, London
  - Moorfields Eye Outreach Unit, St. George's Hospital, London
  - St. Thomas' Hospital, London
  - Oxford Eye Hospital, Oxford
  - Sunderland Eye Infirmary, Sunderland

REFERENCES:
- [Background] Seal DV, Barry P, Gettinby G, Lees F, Peterson M, Revie CW, Wilhelmus KR; ESCRS Endophthalmitis Study Group. ESCRS study of prophylaxis of postoperative endophthalmitis after cataract surgery: Case for a European multicenter study. J Cataract Refract Surg. 2006 Mar;32(3):396-406. doi: 10.1016/j.jcrs.2006.02.014. PMID 16631046
- [Result] Barry P, Seal DV, Gettinby G, Lees F, Peterson M, Revie CW; ESCRS Endophthalmitis Study Group. ESCRS study of prophylaxis of postoperative endophthalmitis after cataract surgery: Preliminary report of principal results from a European multicenter study. J Cataract Refract Surg. 2006 Mar;32(3):407-10. doi: 10.1016/j.jcrs.2006.02.021. PMID 16631047
- [Result] Endophthalmitis Study Group, European Society of Cataract & Refractive Surgeons. Prophylaxis of postoperative endophthalmitis following cataract surgery: results of the ESCRS multicenter study and identification of risk factors. J Cataract Refract Surg. 2007 Jun;33(6):978-88. doi: 10.1016/j.jcrs.2007.02.032. PMID 17531690